CLINICAL TRIAL: NCT05120076
Title: Perioperative Dexamethasone Reduces Postoperative Pain and Nausea After Periacetabular Osteotomy- a Double-blinded Placebo Controlled RCT
Brief Title: Perioperative Dexamethasone Reduces Postoperative Pain and Nausea After Periacetabular Osteotomy
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Balgrist University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DEXA and PAO
Record Dates: First submitted 2021-07-20; First posted 2021-11-15 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Pain; Postoperative Nausea; Amount of Postoperative Opioid Use in Milligrams
MeSH Terms: conditions — Pain; Postoperative Nausea and Vomiting | interventions — Dexamethasone; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Only the investigators as well as the head of anasthesiology will be informed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dexamethasone group (Active Comparator): The patients in the dexamethasone group will receive 12mg dexamethasone (Fortecortin ®) intravenously 15-60 minutes prior to surgery while in general anasthesia as well as 12mg dexamethasone intravenously (Fortecortin®) on the first postoperative day at approx. 8.00a.m. by the investigators.
  Interventions: Drug: Dexamethasone 4 Mg/mL Injectable Solution
- Placebo/ Control group (Placebo Comparator): The patients will not receive any additional drugs preoperatively. 3ml of a 0.9% NaCl Solution (NaCl B. Braun Inf Lös 0.9 % 250ml Ecoflac plus®) will be administered at approx. 8.00 a.m. on the first postoperative day by the investigators.
  Interventions: Drug: NaCl 0.9%

INTERVENTIONS:
Drug: Dexamethasone 4 Mg/mL Injectable Solution — s. arm/group description
  Other Names: Fortecortin Inject (Merck (Switzerland))
  Arms: Dexamethasone group
Drug: NaCl 0.9% — s. arm/group description
  Other Names: NaCL Braun (B Braun medical)
  Arms: Placebo/ Control group

SUMMARY:
The purpose of this study is to assess the effect of Dexamethasone on postoperative pain and nausea after periacetabular osteotomy.

DETAILED DESCRIPTION:
Bernese periacetabular osteotomy (PAO) is a standard procedure with good mid and long-term results. Postoperative pain is a great concern and postoperative pain management of great importance. High demand for opiates and the associated side effects especially nausea limit the postoperative rehabilitation.

Promising results to reduce postoperative pain and nausea have been achieved by perioperative dexamethasone, which has a strong anti-inflammatory effect reducing pain and inflammation as well as a strong anti-emetic effect, especially in total hip replacement.

It is our goal to compare the effect of perioperative intravenous dexamethasone (3x 4mg Amp. Fortecortin =12mg prior to surgery and 3x4mg Amp. Fortecortin = 12mg at 8.00am of the first postoperative day) to a control group (placebo) (3ml saline solution postoperative day 1 at 8.00am) regarding pain level, opiate consumption, postoperative nausea and patient satisfaction.

A double-blinded prospective randomized control trial including up to 60 patients receiving elective unilateral PAO will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* General anasthesia
* Elective periacetabular osteotomy for any reason
* Written informed consent as documented by signature (Appendix Informed Consent Form)
* Competent German language skills

Exclusion Criteria:

* Chronic pain patient, chronic lower back pain
* Steroid or immunosuppressive drugs used within 6 months of surgery
* Renal failure, hepatic failure
* Relevant allergies
* Pregnancy/ Breast feeding
* Contraindications for Fortecortin treatment according to Swissmedic
* Previous enrollment into the current study
* Participation in another study with investigational drug within the 30 days preceding and during the present study
* Known or suspected non-compliance, drug or alcohol abuse Illness according to "Warnings and Precautions of Dexamethasone and NaCl"

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-07-16 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain level | 6 hours postoperatively
  The VAS Pain score assesses pain Levels on a scale from 0 (no pain) to 10 (worst possible pain).
Postoperative pain level | 24 hours postoperatively
  The VAS Pain score assesses pain Levels on a scale from 0 (no pain) to 10 (worst possible pain).
Amount of opiates (morphinequivalent) consumed | 48 hours postoperatively
  The authors will assess the amount of Opiates the Patient needed due to the performed Surgery during the hospital stay.
Amount of anti-emetics consumed (Ondansetron) | 48 hours postoperatively
  The authors will assess the amount of mg of anti- emetic drugs (Ondansetron) the Patient required during the Hospital stay.

SECONDARY OUTCOMES:
Patient satisfaction as assessed by the revised American pain society patient outcome questionnaire | 6 hours postoperatively
  Patient satisfaction will be assessed by the revised American pain Society Patient Outcome questionnaire (APS-POQ-R). (0% worst, 100% best)
Patient satisfaction as assessed by the revised American pain society patient outcome questionnaire | 24 hours postoperatively
  Patient satisfaction will be assessed by the revised American pain Society Patient Outcome questionnaire (APS-POQ-R).(0% worst, 100% best)
Patient satisfaction as assessed by the revised American pain society patient outcome questionnaire | 48 hours postoperatively
  Patient satisfaction will be assessed by the revised American pain Society Patient Outcome questionnaire (APS-POQ-R).(0% worst, 100% best)
Number of vomiting events | 48 hours postoperatively
  The authors will count the number of vomiting events postoperatively as a direct marker for postoperative Nausea.
Physical therapy milestones 1 | 1 week postoperatively
  First steps in the hallway
Physical therapy milestones 2 | 1 week postoperatively
  Walk up stairs
Physical therapy milestones 3 | 1 week postoperatively
  Bicycle ergometer can be used indipendently by the patient
Length of hospitalization | 2 weeks
  The length of hospitalization will be obtained from the Patient Chart.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Zingg, MD, Principal Investigator — Study Principal Investigator
Locations (1):
- Uniklinik Balgrist, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No
No If requested the individual participant data will be made available to other researchers.